CLINICAL TRIAL: NCT02791321
Title: Fragility Assessment in Adults With ADHD and Mental Retardation, Advancing Age
Brief Title: Fragility Assessment in Adults With ADHD and Mental Retardation
Acronym: EFAAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9691
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder; Mental Retardation
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability | interventions — Psychiatry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with ADS-MR (Other): Patients presenting Autism Spectrum Disorder and mental retardation who are evaluated for their ADS severity, their adaptative and intellectual functioning, psychiatric and somatic comorbidities
  Interventions: Other: ADS severity; Other: Adaptative and intellectual functioning; Other: Psychiatric and somatic comorbidities

INTERVENTIONS:
Other: ADS severity — Evaluation of the ADS severity with the CARS scale
Other: Adaptative and intellectual functioning — Evaluation with IQ and Vineland II scale
Other: Psychiatric and somatic comorbidities — Evaluation with the Reiss, DSQIID and CIRS Scales

SUMMARY:
Frailty is a age dependent physiological state of vulnerability. Frailty is screened by the phenotypic model (5 clinical criteria) or the cumulative model (various clinical and biological criteria). Currently, aging with autism spectrum disorder and mental retardation (ADS-MR) is poor described. Nevertheless many data indicate that people with ADS-MR may present an early aging.

Principal aim of this study is to determine if frailty in people with ADS-MR aged over 20 years depend on age. Secondary aims are to evaluate frailty prevalence, to describe with details health according to age, and to verify the frailty index validity for predicting falls, hospitalisation and death, in this population of ADS-MR patients aged over 20 years.

This monocentric and prospective study will include 60 ADS-MR patients aged over 20 years and living in Languedoc-Roussillon's medico-social care homes. Patients are evaluated at the time of inclusion. Frailty index is calculated from 104 clinical and biological criteria. Furthermore the investigator staff collect data about ADS severity (CARS), adaptative and intellectual functionning (Vineland), and psychiatric and somatic comorbidities (Reiss scale, DSQIID and CIRS). Falls, hospitalisations or death occurrence is then collected every year during 5 years.

The connection between frailty index and age will be studied using linear regression. The frailty index validity will be analysed using ROC curves. Modelisation of the falls, hospitalisations or death risk in the 5 years after the initial evaluation will help in identification of the more frailty predictive criteria.

DETAILED DESCRIPTION:
Calendar :

This study will take place during 60 months. 4 first months will be devoted at the ethic and administrative issues. Inclusion will take place during 26 months. Follow-up will take 5 years. Last months will be used for data analysis and articles submission.

Perspectives :

This study will be the first describing frailty evolution during aging in patients suffering from ADS-MR. It will be useful for creating a new, simple and pragmatical frailty screening tool specific for ADS-MR patients in order to detect earlier which patient are the most frail.

ELIGIBILITY:
Inclusion Criteria:

* ADS diagnosis using DSM-5 or CIM-10 criteria, associated to mental retardation
* Age over 20 years
* Patient living in Languedoc-Roussillon's medico-social care home
* Patient benefiting from social security
* Patient or legal representative consent collected

Exclusion criteria:

* Patient or legal representative disagreement to participate at the sudy
* Pregnant woman or nursong mother
* Patient with Down syndrom

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Frailty index | 1 day
  this correspond to the frailty cumulative model : 104 clinical and biological criteria are collected. IF = patient criteria (quoted +1 or 0) sum / evaluated criteria total sum

CONTACTS AND LOCATIONS:
Overall Officials: Amaria BAGHDADLI, PU-PH, Principal Investigator — CRA Peyre Plantade - La Colombière - CHU Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No